CLINICAL TRIAL: NCT04850456
Title: Treatment Strategy of Human Gamma Globulin in Children With Severe Infection Complicated With Inflammatory Storm : A Cohort Study
Brief Title: Treatment Strategy of Human Gamma Globulin on the Therapy for Intensively Ill Children With Inflammatory Storm
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-16
Record Dates: First submitted 2021-03-26; First posted 2021-04-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Critical Illness; Sepsis, Severe
Keywords: Sepsis; Critical Illness; Inflammatory Storm; Gamma Globulin
MeSH Terms: conditions — Critical Illness; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- trial group: Human Gamma Globulin
- control group: conventional treatment

SUMMARY:
The inflammatory storm in critically ill patients releases cytokines, causing systemic immune damage, which may be an important cause of multiple organ failure and even death. Inflammatory storms exacerbate the deterioration of the disease in those children. Gamma globulin may be an effective option to control inflammatory storms. However, this preliminary result needs to be verified from reliable and representative RCTs. In our study, we conducted a retrospective study on the use of gamma globulin and an unused control group. At present, the indications of IVIG are mainly focused on the neuromuscular system and the blood system. We hope to establish a more appropriate and operable evaluation table for the suitability of gamma globulin for clinical use.

DETAILED DESCRIPTION:
In severe infective patients who survive the initial inflammatory storm, the immune response often evolves toward a state of immunosuppression, which contributes to increased mortality and severe secondary hospital-acquired infections. However, the role of gamma globulin therapy in patients with severe infection including sepsis and septic shock is discussed controversially. We intend to retrospectively analyze the efficacy and application evaluation of gamma globulin in severely infected children hospitalized in the intensive care unit. Clinical and demographic data, as well as treatment outcome will be collected from the electronic health record. It is expected to provide evaluation basis for clinicians to formulate treatment plans and clinical pharmacists for special comments on the clinical use of gamma globulin.

ELIGIBILITY:
Inclusion Criteria:

* children hospitalized in PICU of Children's Hospital of Fudan University
* Children With Severe Infection Complicated With Inflammatory Storm

Exclusion Criteria:

* discharge within 48 hours
* patients without informed consent
* incomplete clinical and demographic data

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children hospitalized in PICU of Children's Hospital of Fudan University from January 2022 to December 2023
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The death rate of children | within 28 days after they discharged from PICU
  The death rate of children in 28 days after their discharged from PICU
length of stay in PICU | up to 28 days
  Time from PICU admission to discharge

SECONDARY OUTCOMES:
CD4+/CD8+ | Within 3 to 15 days after the start of treatment
  levels of peripheral blood subgroup of T lymphocyte (digital form)
C-reactive protein (CRP) | Within 3 to 15 days after the start of treatment
  C-reactive protein (digital form)
IL-2R | Within 3 to 15 days after the start of treatment
  The interleukin-2 receptor (digital form)
TNF-alpha | Within 3 to 15 days after the start of treatment
  Tumor necrosis factor alpha (digital form)
Treg | Within 3 to 15 days after the start of treatment
  levels of peripheral blood subgroup of T lymphocyte (digital form)
IL-6 | Within 3 to 15 days after the start of treatment
  The interleukin-6 (digital form)
IFN-gamma | Within 3 to 15 days after the start of treatment
  Interferon gamma (digital form)
Procalcitonin (digital form) | Within 3 to 15 days after the start of treatment
  Procalcitonin (digital form)
IL-10 | Within 3 to 15 days after the start of treatment
  The interleukin-10 (digital form)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai